CLINICAL TRIAL: NCT01768286
Title: A Phase 3, Multicenter, Randomized, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/GS-5885 Fixed-Dose Combination ± Ribavirin for 12 and 24 Weeks in Treatment-Experienced Subjects With Chronic Genotype 1 HCV Infection
Brief Title: Safety and Efficacy of Ledipasvir/Sofosbuvir Fixed-Dose Combination ± Ribavirin in Treatment-Experienced Subjects With Genotype 1 HCV Infection
Acronym: ION-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-337-0109
Record Dates: First submitted 2013-01-10; First posted 2013-01-15 (Estimated); Results first posted 2014-11-26 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2014-11

CONDITIONS: Chronic Hepatitis C Virus
Keywords: HCV genotype 1 (GT-1); HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; GS-7977; GS-5885; Ribavirin; Open Label; Sofosbuvir; Additional relevant MeSH terms:; Hepatitis; Hepatitis, Chronic; Hepatitis C; Hepatitis C, Chronic; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections; Antiviral Agents; Anti-Infective Agents; Therapeutic Uses; Pharmacologic Actions; Antimetabolites; Molecular Mechanisms of Pharmacological Action
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis; Hepatitis, Chronic; Hepatitis C; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- LDV/SOF 12 Weeks (Experimental): Participants will receive LDV/SOF FDC for 12 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 12 Weeks (Experimental): Participants will receive LDV/SOF FDC plus RBV for 12 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV
- LDV/SOF 24 Weeks (Experimental): Participants will receive LDV/SOF FDC for 24 weeks.
  Interventions: Drug: LDV/SOF
- LDV/SOF+RBV 24 Weeks (Experimental): Participants will receive LDV/SOF FDC plus RBV for 24 weeks.
  Interventions: Drug: LDV/SOF; Drug: RBV

INTERVENTIONS:
Drug: LDV/SOF — Ledipasvir (LDV) 90 mg/sofosbuvir (SOF) 400 mg fixed-dose combination (FDC) tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7997
Drug: RBV — Ribavirin (RBV) tablets administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Arms: LDV/SOF+RBV 12 Weeks; LDV/SOF+RBV 24 Weeks

SUMMARY:
This study is to evaluate the safety, tolerability, and antiviral efficacy of ledipasvir/sofosbuvir fixed dose combination (FDC) with or without ribavirin (RBV) administered for 12 or 24 weeks in treatment-experienced subjects with chronic genotype 1 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18, with chronic genotype 1 HCV infection
* HCV treatment-experienced, including patients who have previously failed a nonstructural protein (NS)3/4A protease inhibitor plus pegylated interferon (PEG)/RBV regimen
* HCV RNA > 10,000 IU/mL at screening
* Cirrhosis determination; a liver biopsy may be required
* Screening laboratory values within defined thresholds
* Use of two effective contraception methods if female of childbearing potential or sexually active male

Exclusion Criteria:

* Pregnant or nursing female or male with pregnant female partner
* Coinfection with HIV or hepatitis B virus
* Current or prior history of clinical hepatic decompensation
* Hepatocellular carcinoma or other malignancy (with exception of certain resolved skin cancers)
* Chronic use of systemic immunosuppressive agents
* History of clinically significant illness or any other medical disorder that may interfere with subject treatment, assessment or compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2013-01; Primary Completion 2013-11 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Yang, PharmD, Study Director — Gilead Sciences
Locations (53):
- United States (53):
  - Phoenix, Arizona
  - Tucson, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Palo Alto, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Englewood, Colorado
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Bowling Green, Kentucky
  - Baton Rouge, Louisiana
  - Baltimore, Maryland
  - Lutherville, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Rochester, Minnesota
  - Saint Louis, Minnesota
  - Saint Paul, Minnesota
  - Kansas City, Missouri
  - Berlin, New Jersey
  - Hillsborough, New Jersey
  - Albuquerque, New Mexico
  - Santa Fe, New Mexico
  - Binghamton, New York
  - Manhasset, New York
  - New York, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Fayetteville, North Carolina
  - Statesville, North Carolina
  - Winston-Salem, North Carolina
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Newport News, Virginia
  - Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

REFERENCES:
- [Derived] Grebely J, Mauss S, Brown A, Bronowicki JP, Puoti M, Wyles D, Natha M, Zhu Y, Yang J, Kreter B, Brainard DM, Yun C, Carr V, Dore GJ. Efficacy and Safety of Ledipasvir/Sofosbuvir With and Without Ribavirin in Patients With Chronic HCV Genotype 1 Infection Receiving Opioid Substitution Therapy: Analysis of Phase 3 ION Trials. Clin Infect Dis. 2016 Dec 1;63(11):1405-1411. doi: 10.1093/cid/ciw580. Epub 2016 Aug 23. PMID 27553375
- [Derived] Afdhal N, Reddy KR, Nelson DR, Lawitz E, Gordon SC, Schiff E, Nahass R, Ghalib R, Gitlin N, Herring R, Lalezari J, Younes ZH, Pockros PJ, Di Bisceglie AM, Arora S, Subramanian GM, Zhu Y, Dvory-Sobol H, Yang JC, Pang PS, Symonds WT, McHutchison JG, Muir AJ, Sulkowski M, Kwo P; ION-2 Investigators. Ledipasvir and sofosbuvir for previously treated HCV genotype 1 infection. N Engl J Med. 2014 Apr 17;370(16):1483-93. doi: 10.1056/NEJMoa1316366. Epub 2014 Apr 11. PMID 24725238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 64 study sites in the United States. The first participant was screened on 03 January 2013. The last participant observation occurred on 20 February 2014.
Pre-assignment Details: 551 participants were screened.
Groups:
- LDV/SOF 12 Weeks: Ledipasvir (LDV) 90 mg/sofosbuvir (SOF) 400 mg fixed-dose combination (FDC) tablet once daily for 12 weeks
- LDV/SOF+RBV 12 Weeks: LDV 90 mg/SOF 400 mg FDC tablet once daily plus ribavirin (RBV) tablets (1000-1200 mg daily based on weight) for 12 weeks
- LDV/SOF 24 Weeks: LDV 90 mg/SOF 400 mg FDC tablet once daily for 24 weeks
- LDV/SOF+RBV 24 Weeks: LDV 90 mg/SOF 400 mg FDC tablet once daily plus RBV tablets (1000-1200 mg daily based on weight) for 24 weeks
Period: Overall Study
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Started | 109 | 111 | 110 | 111
Completed | 102 | 107 | 108 | 110
Not Completed | 7 | 4 | 2 | 1
Not completed — Randomized But Not Treated | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 7 | 4 | 0 | 1
Not completed — Withdrew Consent | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were randomized and received at least one dose of study drug. Participants failed a previous HCV treatment regimen consisting of pegylated interferon alfa-2a (Pegasys) or pegylated interferon alfa-2b (Pegintron) plus ribavirin (RBV), with or without a protease inhibitor (PI).
Groups:
- LDV/SOF 12 Weeks: LDV 90 mg/SOF 400 mg FDC tablet once daily for 12 weeks
- LDV/SOF+RBV 12 Weeks: LDV 90 mg/SOF 400 mg FDC tablet once daily plus RBV tablets (1000-1200 mg daily based on weight) for 12 weeks
- Total: Total of all reporting groups
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks | Total
Number analyzed (Participants) | 109 | 111 | 109 | 111 | 440
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (6.9) | 57 (8.0) | 56 (8.3) | 55 (7.8) | 56 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 40 | 35 | 43 | 153
  Male | 74 | 71 | 74 | 68 | 287
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 24 | 16 | 17 | 20 | 77
  White | 84 | 94 | 91 | 89 | 358
  Asian | 1 | 0 | 0 | 0 | 1
  Hawaiian or Pacific Islander | 0 | 1 | 0 | 1 | 2
  Other | 0 | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic/Latino | 7 | 12 | 11 | 11 | 41
  Not Hispanic or Latino | 100 | 99 | 98 | 99 | 396
  Not Disclosed | 2 | 0 | 0 | 1 | 3
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.5 (0.44) | 6.4 (0.54) | 6.4 (0.57) | 6.5 (0.60) | 6.5 (0.54)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 6 | 13 | 16 | 15 | 50
  ≥ 800,000 IU/mL | 103 | 98 | 93 | 96 | 390
HCV Genotype [Number; unit: participants]
  Genotype 1a | 86 | 88 | 85 | 88 | 347
  Genotype 1b | 23 | 23 | 24 | 23 | 93
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 10 | 11 | 16 | 18 | 55
    CT | 70 | 77 | 68 | 68 | 283
    TT | 29 | 23 | 25 | 25 | 102
Prior HCV Treatment [Number; unit: participants] — IFN-alfa-2b = interferon-alfa 2b; PEG-IFN-alfa-2a = pegylated interferon alfa-2a; PEG-IFN-alfa-2b - pegylated interferon alfa-2b; RBV = ribavirin; PI = protease inhibitor
  participants
    PEG-IFN-alfa-2a or PEG-IFN-alfa-2b+RBV | 43 | 47 | 58 | 59 | 207
    PI+PEG-IFN-alfa-2a or PEG-IFN-alfa-2b+RBV | 66 | 64 | 50 | 51 | 231
    IFN-alfa-2b+RBV | 0 | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) 12 weeks following the last dose of study drug.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants who were randomized and received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 111
percentage of participants | 93.6 | 96.4 | 99.1 | 99.1
Statistical Analysis 1: Comparison: LDV/SOF 12 Weeks; Test type: Superiority or Other; p < 0.001, Binomial test — A 2-sided 1-sample binomial test was used to compare over the historical SVR12 rate of 25%. To control the family-wise type I error rate at 0.05, the Hochberg procedure was applied, from which the adjusted p-values were obtained
Statistical Analysis 2: Comparison: LDV/SOF+RBV 12 Weeks; Test type: Superiority or Other; p < 0.001, Binomial test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: LDV/SOF 24 Weeks; Test type: Superiority or Other; p < 0.001, Binomial test — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: LDV/SOF+RBV 24 Weeks; Test type: Superiority or Other; p < 0.001, Binomial test — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Incidence of Adverse Events Leading to Permanent Discontinuation From Any Study Drug
Description: The percentage of participants who experienced an adverse event leading to permanent discontinuation from any study drug was summarized.
Time Frame: Up to 24 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 111
percentage of participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With SVR at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 111
percentage of participants
  SVR4 | 94.5 | 96.4 | 100.0 | 99.1
  SVR24 | 93.6 | 96.4 | 99.1 | 99.1

4. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 1
Time Frame: Week 1
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 111
percentage of participants | 26.6 | 33.3 | 20.2 | 29.7

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 2
Time Frame: Week 2
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 111
percentage of participants | 81.7 | 82.9 | 81.7 | 83.8

6. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 4
Time Frame: Week 4
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 111
percentage of participants | 100.0 | 99.1 | 99.1 | 99.1

7. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 8
Time Frame: Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 110
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0

8. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 12
Time Frame: Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 110
percentage of participants | 99.1 | 100.0 | 100.0 | 100.0

9. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ at Week 24
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed. Participants in the LDV/SOF 12 Weeks and LDV/SOF+RBV 12 Weeks groups did not continue treatment past Week 12 and are not included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 0 | 0 | 107 | 110
percentage of participants |  |  | 100.0 | 100.0

10. Secondary Outcome: Change From Baseline in HCV RNA at Week 1
Time Frame: Baseline; Week 1
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 108 | 111 | 109 | 110
log10 IU/mL | -4.57 (0.501) | -4.50 (0.540) | -4.47 (0.569) | -4.50 (0.575)

11. Secondary Outcome: Change From Baseline in HCV RNA at Week 2
Time Frame: Baseline; Week 2
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 111
log10 IU/mL | -5.08 (0.443) | -4.94 (0.520) | -4.99 (0.571) | -4.99 (0.617)

12. Secondary Outcome: Change From Baseline in HCV RNA at Week 4
Time Frame: Baseline; Week 4
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 111
log10 IU/mL | -5.16 (0.439) | -5.02 (0.543) | -5.06 (0.571) | -5.04 (0.779)

13. Secondary Outcome: Change From Baseline in HCV RNA at Week 8
Time Frame: Baseline; Week 8
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 110
log10 IU/mL | -5.16 (0.439) | -5.02 (0.544) | -5.06 (0.571) | -5.08 (0.605)

14. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as on-treatment virologic failure or virologic relapse.
  * On-Treatment Virologic Failure was defined as
    * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
    * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
    * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
  Virologic relapse was defined as confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Baseline to posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Number analyzed (Participants) | 109 | 111 | 109 | 111
percentage of participants
  On-Treatment Virologic Failure | 0 | 0 | 0 | 0.9
  Virologic relapse | 6.5 | 3.6 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | LDV/SOF 12 Weeks | LDV/SOF+RBV 12 Weeks | LDV/SOF 24 Weeks | LDV/SOF+RBV 24 Weeks
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/111 | 6/109 | 3/111
Other Adverse Events (participants affected / at risk) | 73/109 | 96/111 | 87/109 | 100/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (N=109) | LDV/SOF+RBV 12 Weeks (N=111) | LDV/SOF 24 Weeks (N=109) | LDV/SOF+RBV 24 Weeks (N=111)
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF 12 Weeks (N=109) | LDV/SOF+RBV 12 Weeks (N=111) | LDV/SOF 24 Weeks (N=109) | LDV/SOF+RBV 24 Weeks (N=111)
Anaemia (Blood and lymphatic system disorders) | 0 | 9 | 1 | 12
Nausea (Gastrointestinal disorders) | 13 | 20 | 7 | 25
Diarrhoea (Gastrointestinal disorders) | 7 | 5 | 9 | 17
Constipation (Gastrointestinal disorders) | 2 | 4 | 6 | 3
Vomiting (Gastrointestinal disorders) | 2 | 3 | 0 | 9
Abdominal pain (Gastrointestinal disorders) | 6 | 2 | 0 | 5
Fatigue (General disorders) | 23 | 45 | 26 | 50
Irritability (General disorders) | 2 | 13 | 4 | 12
Upper respiratory tract infection (Infections and infestations) | 4 | 6 | 7 | 11
Bronchitis (Infections and infestations) | 2 | 3 | 4 | 8
Nasopharyngitis (Infections and infestations) | 3 | 5 | 3 | 6
Sinusitis (Infections and infestations) | 1 | 6 | 3 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 13 | 7 | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 6 | 8 | 10
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 8 | 2 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 4 | 10
Headache (Nervous system disorders) | 28 | 26 | 25 | 35
Dizziness (Nervous system disorders) | 3 | 8 | 7 | 12
Insomnia (Psychiatric disorders) | 10 | 18 | 4 | 19
Anxiety (Psychiatric disorders) | 2 | 7 | 4 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 16 | 5 | 16
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 16 | 3 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 6
Rash (Skin and subcutaneous tissue disorders) | 2 | 11 | 6 | 16
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 10 | 2 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years